CLINICAL TRIAL: NCT00081302
Title: A Phase II Study Of Cetuximab (C225) In Combination With Chemoradiation In Patients With Stage IIIA/B Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Cetuximab, Paclitaxel, Carboplatin, and Radiation Therapy in Treating Patients With Unresectable Stage IIIA or Stage IIIB Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: RTOG-0324; CDR0000352163
Record Dates: First submitted 2004-04-07; First posted 2004-04-08 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Lung Cancer
Keywords: stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; squamous cell lung cancer; large cell lung cancer; adenocarcinoma of the lung; bronchoalveolar cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar | interventions — Cetuximab; Carboplatin; Paclitaxel; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: cetuximab
Drug: carboplatin
Drug: paclitaxel
Radiation: radiation therapy

SUMMARY:
RATIONALE: Monoclonal antibodies such as cetuximab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Drugs used in chemotherapy, such as paclitaxel and carboplatin, work in different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Giving cetuximab together with combination chemotherapy and radiation therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving cetuximab together with paclitaxel, carboplatin, and radiation therapy works in treating patients with unresectable stage IIIA or stage IIIB non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the feasibility of cetuximab when administered concurrently with paclitaxel, carboplatin, and radiotherapy, in terms of safety and compliance, in patients with unresectable stage IIIA or IIIB non-small cell lung cancer.

Secondary

* Determine the response rate (complete and partial) in patients treated with this regimen.
* Determine the overall survival (1- and 2-year survival rate and median survival) of patients treated with this regimen.
* Determine the time to disease progression (at 1 and 2 years) in patients treated with this regimen.
* Correlate epidermal growth factor receptor expression with the toxicity of this regimen and response, overall survival, and progression in these patients.

OUTLINE: This is a multicenter study.

* Cetuximab loading dose (week 1): Patients receive a loading dose of cetuximab IV over 2 hours on day 1.
* Concurrent cetuximab and chemoradiotherapy (weeks 2-8): Patients receive cetuximab IV over 1 hour, paclitaxel IV over 1 hour, and carboplatin IV over 30 minutes on days 8, 15, 22, 29, 36, 43, and 50. Patients undergo radiotherapy once daily on days 8-12, 15-19, 22-26, 29-33, 36-40, 43-47, and 50-53.
* Consolidation therapy (weeks 9-17): Patients receive cetuximab IV over 1 hour on days 57, 64, 71, 78, 85, 92, 99, 106, and 113. Patients also receive paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on days 78 and 99.

Treatment continues in the absence of disease progression or unacceptable toxicity.

Patients are followed at 30 days, every 3 months for 2 years, every 4 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 84 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC) of 1 of the following subtypes:

  * Squamous cell carcinoma
  * Adenocarcinoma (including bronchoalveolar cell)
  * Large cell anaplastic carcinoma (including giant and clear cell carcinomas)
  * Poorly differentiated/not otherwise specified NSCLC
* Stage IIIA (T1-2, N2, M0 or T3, N1-2, M0) or IIIB (T4, any N, M0 or any T, N2-3, M0)

  * If the largest mediastinal node is < 2.0 cm in diameter and this is the basis for stage III disease, then at least 1 of the nodes must be cytologically or histologically positive
* Unresectable disease

  * No totally resected tumors
* Tumors adjacent to a vertebral body allowed provided all gross disease can be encompassed in the radiation boost field and the boost volume is limited to < 50% of the ipsilateral lung volume
* Measurable disease
* Transudate, cytologically negative, non-bloody pleural effusions allowed provided the tumor can be encompassed within a reasonable field of radiotherapy

  * Pleural effusions seen on a chest CT scan are allowed provided they are not visible on a chest x-ray and are too small to tap
* No asymptomatic or symptomatic brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Zubrod 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9 g/dL (transfusion independent)

Hepatic

* Bilirubin ≤ 1.5 mg/dL
* SGOT (serum glutamic oxaloacetic transaminase) or SGPT (serum glutamate pyruvate transaminase) ≤ 3 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2.5 times ULN

Renal

* Creatinine ≤ 2.0 mg/dL

Cardiovascular

* No significant history of cardiac disease
* No uncontrolled hypertension
* No unstable angina
* No uncompensated congestive heart failure
* No myocardial infarction within the past year
* No cardiac ventricular arrhythmias requiring medication
* LVEF (left ventricular ejection fraction) normal by MUGA (multi-gated acquisition) scan or echocardiogram

Pulmonary

* No history of interstitial pneumonitis
* No history of severe chronic obstructive pulmonary disease requiring 3 or more hospitalizations within the past year
* FEV_1 ≥ 1,200 cc
* No active pulmonary infection unresponsive to conventional antibiotics

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 4 weeks after study therapy
* Glucose ≤ 2 times ULN
* No more than 5% weight loss within the past 3 months
* No known allergy to murine proteins or Cremophor EL
* No neuropathy grade 2 or greater
* No other malignancy within the past 2 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or other in situ cancers

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior drugs that target the epidermal growth factor receptor pathway
* No prior chimerized monoclonal antibody therapy
* No other concurrent immunotherapy
* No concurrent colony-stimulating factors (i.e., filgrastim [G-CSF] and sargramostim [GM-CSF])

  * Concurrent epoetin alfa allowed

Chemotherapy

* No prior systemic chemotherapy
* No other concurrent chemotherapy

Endocrine therapy

* No concurrent hormonal therapy except hormones for non-disease-related conditions (e.g., insulin for diabetes) or steroids for acute symptom management, adrenal failure, septic shock, or as antiemetics

Radiotherapy

* No prior thoracic or neck radiotherapy
* No concurrent intensity-modulated radiotherapy

Surgery

* Recovered from prior exploratory thoracotomy
* No prior surgical resection of the present cancer

Other

* More than 30 days since prior participation in another clinical trial
* No concurrent participation in another clinical trial
* No other concurrent anticancer therapy
* No amifostine during or for 3 months after study radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-03; Primary Completion 2005-12 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George R. Blumenschein, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- Arlington Cancer Center - Arlington, Arlington, Texas, United States

REFERENCES:
- [Result] Blumenschein GR Jr, Paulus R, Curran WJ, Robert F, Fossella F, Werner-Wasik M, Herbst RS, Doescher PO, Choy H, Komaki R. Phase II study of cetuximab in combination with chemoradiation in patients with stage IIIA/B non-small-cell lung cancer: RTOG 0324. J Clin Oncol. 2011 Jun 10;29(17):2312-8. doi: 10.1200/JCO.2010.31.7875. Epub 2011 May 9. PMID 21555682
- [Result] Blumenschein GR, Paulus R, Curran WJ, et al.: A phase II study of cetuximab (C225) in combination with chemoradiation (CRT) in patients (PTS) with stage IIIA/B non-small cell lung cancer (NSCLC): A report of the 2 year and median survival (MS) for the RTOG 0324 trial. [Abstract] J Clin Oncol 26 (Suppl 15): A-7516, 2008.
- [Result] Olsen CC, Paulus R, Komaki R, et al.: RTOG 0324: A phase II study of cetuximab (C225) in combination with chemoradiation (CRT) in patients with stage IIIA/B non-small cell lung cancer (NSCLC)--Association between EGFR gene copy number and patients' outcome. [Abstract] J Clin Oncol 26 (Suppl 15): A-7607, 2008.
- [Result] Blumenschein G Jr, Moughan J, Curran W, et al.: A phase II study of cetuximab (C225) in combination with chemoradiation (CRT) in patients (pts) with stage III A/B non-small cell lung cancer (NSCLC): an interim report of the RTOG 0324 trial. [Abstract] J Clin Oncol 25 (Suppl 18): A-7531, 392s, 2007.
- [Result] Komaki R, Moughan J, Ang K, et al.: RTOG 0324: a phase II study of cetuximab (C225) in combination with chemoradiation (CRT) in patients (PTS) with stage IIIA/B non-small cell lung cancer (NSCLC): correlation between EGFR expression and the patients' outcome. [Abstract] Int J Radiat Oncol Biol Phys 69 (3 Suppl): A-101, S57-58, 2007.
- [Result] Werner-Wasik M, Swann S, Curran W, et al.: A phase II study of cetuximab (C225) in combination with chemoradiation (CRT) in patients (PTS) with stage IIIA/B non-small cell lung cancer (NSCLC): an interim overall toxicity report of the RTOG 0324 trial. [Abstract] J Clin Oncol 23 (Suppl 16): A-7135, 654s, 2005.